CLINICAL TRIAL: NCT04303962
Title: An Observational Cohort Study on the Efficacy of Intravenous Gamma Globulin on Guillain-Barre Syndrome
Brief Title: Efficacy of Intravenous Gamma Globulin on Guillain-Barre Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Director, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA，ECFAH of FMU[2019]217
Record Dates: First submitted 2020-02-28; First posted 2020-03-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Guillain-barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Guillain-barre syndrome (GBS) is an acute immune-mediated polyneuropathy. Intravenous Gamma globulin is an effective therapy.Although high doses of gamma globulin are clinically effective, the patient's recovery and clinical prognosis vary. The establishment of a cohort study on the therapeutic effect of gamma globulin in Guillain-barre Syndrome is beneficial to the diagnosis of the disease and to the understanding of the natural course of the disease and the efficacy of drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Brighton Guillain-Barre Syndrome diagnosis criteria in 2014;
2. Age ≥18;
3. Patients with AIDP, AMAN and AMSAN;

5. IVIG was treated within 2 weeks of onset; 6. GBS disability scale>2; 6. Cooperate with patients who were followed up for 180 days and sign the informed consent;

Exclusion criteria:

1. Age <18;
2. Pregnant or nursing women;
3. Patients with Chronic inflammatory demyelinating multiple peripheral neuropathy;
4. Combined with other types of immune system diseases;
5. Accept drugs that affect the function of the immune system within 5 or 3 months;
6. Concomitant neoplastic diseases.
7. The patient or guardian refused to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with GBS after standard IVIg treatment in relation to slow clinical course or worse outcome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
GBS disability score | 6 months
  GBS disability scale ( Guillain-Barré syndrome disability scale) was defined as follows: 0: healthy state; 1: minor symptoms and capable of running; 2: able to walk 5 meters or more without assistance but unable to run; 3: able to walk 5 meters across an open space with help; 4: bedridden or chair-bound; 5: requiring assisted ventilation for at least part of the day; 6: dead

SECONDARY OUTCOMES:
Respiratory function | 6 months
  whether mechanical ventilation is required

CONTACTS AND LOCATIONS:
Overall Officials: Ning Wang, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Neurology,First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China